CLINICAL TRIAL: NCT01216202
Title: Sexual Function and Wellbeing in Males Diagnosed With Rectal Cancer
Brief Title: Sexual Function and Wellbeing in Males With Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Cancer Society (Other)
Responsible Party: Principal Investigator, Anna Martling, Professor, Senior Consultant Surgeon, Karolinska Institutet
Other Study IDs: 2009/1860-31/2
Record Dates: First submitted 2010-10-04; First posted 2010-10-07 (Estimated); Results first posted 2021-04-02 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Preoperative radiotherapy; Pelvic surgery; Sexual function; Wellbeing; Hormone levels; Spermatogenesis
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood- and semen samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Preoperative RT: Men with rectal cancer treated with preoperative radiotherapy (RT) and surgery.
  Interventions: Radiation: Preoperative radiotherapy
- No preoperative RT: Men with rectal cancer or prostate cancer treated with surgery alone (no RT).

INTERVENTIONS:
Radiation: Preoperative radiotherapy — Preoperative radiotherapy (RT) was administered as either short course (5Gy x5) or long-course (2Gy x25 or 1.8 Gy x25 with or without 3 fractions of boost to the primary tumor and radiologically malignant lymph nodes) treatment with or without concomitant or sequential chemotherapy. Oncological treatment was decided at a multidisciplinary team conference.
  Testicular doses (TDs) was calculated from planning CT-scans and reported as mean cumulative testicular dose. Relative TD was calculated based in the assumption that RT regimens for rectal cancer are bioequivalent and referred to as proportion of prescribed dose absorbed by the testes.
  Groups: Preoperative RT

SUMMARY:
Preoperative radiotherapy and pelvic surgery is recommended to many patients with rectal cancer. For men there are theoretical reasons to believe that the treatment may effect hormone levels, spermatogenesis, sexual function and wellbeing. To address these questions a longitudinal observational study was initiated where measurements of androgen hormone levels, semen samples and sexual function were assessed before treatment (baseline) and during a follow-up period of two years.

DETAILED DESCRIPTION:
Men with rectal cancer stage I to III planned for resection was included in the study. Men treated with preoperative RT were assigned to the exposed group and men treated with surgery alone were assigned to the unexposed group. Eighteen months after start of inclusion, less than 10% of the participants were treated with surgery alone. To increase the sample size of the unexposed group, men with prostate cancer stage I to III and scheduled for robot-assisted prostatectomy were also included.

Participants with rectal cancer were enrolled at two centres in Stockholm (Karolinska University Hospital and Ersta Hospital) between 2010 and 2014. Participants with prostate cancer were enrolled at the Urology department of the Karolinska University Hospital in Stockholm between 2012 and 2013.

Patient data, fasting venous blood samples, semen samples and questionnaires regarding sexual function and well being were collected before start of oncological treatment (baseline), 1 and 2 years after surgery. Men treated with preoperative RT for rectal cancer had an additional venous blood sample during the week before surgery. Men with rectal cancer under 55 years of age were offered semen cryopreservation.

Participants could choose if they wanted to participate in one, two or three of the following parts; hormone analysis, semen analysis and/ or questionnaires regarding sexual function and well being. Semen sampling and cryopreservation was not performed in men with prostate cancer.

Changes in hormone levels, semen measurements and sexual function during follow-up were assessed, and compared between exposed and unexposed participants.

ELIGIBILITY:
Inclusion Criteria:

* Males diagnosed with rectal cancer stadium I-III, planned for surgery with or without preoperative radiotherapy or males with prostate cancer stadium I-III planned for robot-assisted prostatectomy without preoperative radiotherapy.
* Informed consent
* Fluent in Swedish
* Residents of the Stockholm county area

Exclusion Criteria:

* Rectal cancer stadium IV
* Previous radiotherapy to the pelvic region
* History or evidence of a second pelvic malignancy
* Androgen deprivation therapy, Testosterone replacement or Androgen abuse

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with rectal cancer stadium I-III, planned for abdominal surgery with or without preoperative radiotherapy.
  Men with prostate cancer stadium I-III planned for robot-assisted prostatectomy (no preoperative radiotherapy).
Sampling Method: Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2010-04; Primary Completion 2014-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Martling, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Ersta Hospital, Stockholm
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buchli C, Tapper J, Bottai M, Holm T, Arver S, Blomqvist L, Martling A. Testosterone and body composition in men after treatment for rectal cancer. J Sex Med. 2015 Mar;12(3):774-82. doi: 10.1111/jsm.12751. Epub 2014 Nov 12. PMID 25388654
- [Background] Buchli C, Al Abani M, Ahlberg M, Holm T, Fokstuen T, Bottai M, Frodin JE, Lax I, Martling A. Assessment of testicular dose during preoperative radiotherapy for rectal cancer. Acta Oncol. 2016;55(4):496-501. doi: 10.3109/0284186X.2015.1073349. Epub 2015 Sep 11. PMID 26362484
- [Background] Tapper J, Arver S, Holm T, Bottai M, Machado M, Jasuja R, Martling A, Buchli C. Acute primary testicular failure due to radiotherapy increases risk of severe postoperative adverse events in rectal cancer patients. Eur J Surg Oncol. 2020 Jan;46(1):98-104. doi: 10.1016/j.ejso.2019.07.023. Epub 2019 Jul 19. PMID 31350073
- [Result] Buchli C, Martling A, Abani MA, Frodin JE, Bottai M, Lax I, Arver S, Holm T. Risk of Acute Testicular Failure After Preoperative Radiotherapy for Rectal Cancer: A Prospective Cohort Study. Ann Surg. 2018 Feb;267(2):326-331. doi: 10.1097/SLA.0000000000002081. PMID 27849668

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with rectal cancer stage I to III planned for rectal resection eligible for the study were enrolled at a tertiary (Karolinska University Hospital) and secondary hospital (Ersta Hospital) in Stockholm during April 2010 and May 2014. Of 372 men with rectal cancer assessed for eligibility, 115 were included in the study.
Pre-assignment Details: 18 months after start of inclusion, less than 10% of the participants were treated with surgery alone. To increase the sample size of the unexposed group (no preoperative radiotherapy), 63 men with prostate cancer I to III scheduled for robot assisted prostatectomy were included. Participants with prostate cancer were enrolled at the Urology department at Karolinska University Hospital between May 2012 and January 2013.
Period: Overall Study
Arm/Group | Preoperative RT | No Preoperative RT
Started (Included in the study) | 101 | 77
Analysed at Baseline | 93 | 75
Analysed After RT | 79 | 0
Completed (Analysed at baseline) | 79 | 75
Not Completed | 22 | 2
Not completed — Withdrawal by Subject | 8 | 0
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 14 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preoperative RT | No Preoperative RT | Total
Number analyzed (Participants) | 93 | 75 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (11.3) | 63.3 (6.7) | 61.6 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 93 | 75 | 168
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.3 (4.1) | 26.4 (3.0) | 25.8 (3.7)
ASA score [Count of Participants; unit: Participants] — ASA score is a classification system for physical status ranging from scores I to VI with higher scores indicting worse physical status. Definitions of scores; I = Normal healthy person, II = A patient with mild systemic disease, III = A patient with severe systemic disease.
  Participants
    I | 21 | 25 | 46
    II | 51 | 41 | 92
    III | 21 | 7 | 28
    Missing data | 0 | 2 | 2
Preoperative RT [Count of Participants; unit: Participants]
  Short course RT (5x5 Gy) | 68 | 0 | 68
  Long course RT (1.8x28 Gy) | 25 | 0 | 25
  No RT | 0 | 75 | 75
Preoperative chemotherapy [Count of Participants; unit: Participants]
  Concomitant chemotherapy | 23 | 0 | 23
  Full dose chemotherapy | 11 | 0 | 11
  No chemotherapy | 59 | 75 | 134

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Testosterone Levels Between Baseline and After Preoperative Radiotherapy.
Description: Fasting morning venous blood samples were collected at baseline, eg prior to oncological treatment. Men with rectal cancer treated with preoperative radiotherapy (RT) had a second blood sample taken afte RT and before surgery, collected the week before surgery and defined as "after RT/before surgery". Elapsed time between start of RT and the second blood sample was median 38 days, ranging from 3 to 195 days depending on the type of preoperative oncological treatment regimen. Testosterone (T) was analysed at the Department of Clinical Chemistry, Karolinska University Hospital, using commercial assays.
Time Frame: Baseline and after RT/before surgery.
Population: For participants in "No preoperative RT", no blood samples were collected at the time point "after RT/before surgery".
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Preoperative RT | No Preoperative RT
Number analyzed (Participants) | 93 | 75
nmol/L
  Baseline | 11.3 (3.4) | 11.9 (4.0)
  After RT/before surgery: number analyzed (Participants) | 79 | 0
  After RT/before surgery | 9.3 (3.5) |
Statistical Analysis 1: Comparison: Preoperative RT vs No Preoperative RT; The association between change in serum testosterone levels and cumulative mean testicular radiation dose was assessed using longitudinal regression analysis (GEE). No preoperative RT contributed with baseline values; Test type: Superiority; p = 0.014, Regression, Linear — The threshold for statistical significance was p = 0.05

2. Primary Outcome: Change in Total Number of Sperms Per Ejaculate Between Baseline and Two Year Follow-up.
Description: Semen samples were collected at the Department of Reproductive Medicine of Karolinska University Hospital after 72h of sexual abstinence and analysed according to World Health Organization 2010 standard. Total number of sperms (million spermatozoa per ejaculate), was calculated by multiplying sperm concentration (million spermatozoa per millilitre semen) with semen volume (milliliter semen/ejaculate). Total number of sperms below 39 million per ejaculate was defined as oligospermia, and 0 million per ejaculate was defined as azoospermia. Semen samples were only collected in men with rectal cancer, not prostate cancer.
Time Frame: Baseline, 1 and 2 years after surgery.
Population: Of the 115 men with rectal cancer included in the study, 21 men left at least one semen sample during the study period and was included in the analysis. 20 of 21 men had RT. In total 40 semen samples was analysed. During follow-up three participants with RT dropped out of the study. Number analysed at each time points represents number of available semen samples at each time point; 19 of 21 at baseline, 9 of 18 1 year after surgery, 12 of 18 2 year after surgery.
Measure: Median (Full Range); unit: million spermatozoa per ejaculate
Units Other Than Participants: Semen samples
Groups:
- Preoperative RT: Men with rectal cancer treated with preoperative therapy (RT) and surgery with available semen samples.
- No Preoperative RT: Men with rectal cancer treated with surgery alone (no RT) with available semen samples.
Arm/Group | Preoperative RT | No Preoperative RT
Number analyzed (Participants) | 20 | 1
Number analyzed (Semen samples) | 39 | 1
million spermatozoa per ejaculate
  Baseline: number analyzed (Semen samples) | 19 | 0
  Baseline | 164.0 [5.9 to 1140.0] |
  1 year after surgery: number analyzed (Participants) | 17 | 1
  1 year after surgery: number analyzed (Semen samples) | 8 | 1
  1 year after surgery | 3.15 [0.0 to 216.0] | 0.0 [0.0 to 0.0]
  2 years after surgery: number analyzed (Participants) | 17 | 1
  2 years after surgery: number analyzed (Semen samples) | 12 | 0
  2 years after surgery | 32.6 [0.0 to 187.0] |
Statistical Analysis 1: Comparison: Preoperative RT; The association between change in total number of sperms per ejaculate and relative mean testicular dose was assessed using longitudinal regression analysis (GEE); Test type: Superiority; p = 0.008, Regression, Linear — The threshold for statistical significance was p=0.05; Model adjusted for time between preoperative radiotherapy (RT) and surgery; Estimated mean change = -4.0, 95% CI 2-sided [-6.9 to -1.0]

3. Primary Outcome: Sexual Function
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2024-06

ADVERSE EVENTS:
Description: Adverse events were not monitored.
Groups:
- Preoperative RT: Men with rectal cancer treated with preoperative therapy (RT) and surgery.
Arm/Group | Preoperative RT | No Preoperative RT
All-Cause Mortality (participants affected / at risk) | 0/101 | 2/77
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes